CLINICAL TRIAL: NCT07059780
Title: A Randomized Controlled Trial Investigating the Effect of Virtual Reality Glasses on Anxiety and Pain Levels in Women During Gynecological Examination
Brief Title: Effect of Virtual Reality on Anxiety and Pain During Gynecological Examination
Acronym: VR-GYN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fazilet Nur Daşkın (Other)
Responsible Party: Sponsor-Investigator, Fazilet Nur Daşkın, MSc Student in Nursing, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ERU-SBE-FND-2025; 2023/728 (Other: Erciyes University Clinical Research Ethics Committee)
Record Dates: First submitted 2025-06-23; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Pain; Gynecological Examination; Women's Health
Keywords: anxiety; pain; virtual reality; Women's Health; gynecological examination
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to two groups: the intervention group received virtual reality during the procedure, and the control group received standard care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Intervention Group (Experimental): Participants in this group underwent a routine gynecological examination while wearing virtual reality glasses that displayed immersive nature-themed videos with visual and auditory stimuli to reduce anxiety and pain.
  Interventions: Device: Virtual Reality Glasses
- Routine Care Without VR Group (No Intervention): Participants in this group received standard gynecological examination without any virtual reality intervention. No visual or auditory stimulus was provided during the procedure.

INTERVENTIONS:
Device: Virtual Reality Glasses — Participants in the intervention group wore virtual reality (VR) glasses during the gynecological examination. The VR content included immersive nature-themed scenes accompanied by calming background music. The intervention aimed to provide a multisensory distraction to reduce perceived anxiety and pain levels during the procedure.
  Arms: Virtual Reality Intervention Group

SUMMARY:
This randomized controlled trial aims to examine the effects of using virtual reality (VR) glasses during gynecological examinations on women's pain and anxiety levels. A total of 126 women were randomly assigned to either an intervention group, who used VR glasses during the examination, or a control group, who received standard care. Visual and auditory stimuli from nature-themed videos were shown to the intervention group using VR glasses during the procedure. Participants' pain was assessed using the Visual Analog Scale (VAS), and anxiety was measured using the State-Trait Anxiety Inventory (STAI-I). The study was conducted between February and November 2024 at the Department of Obstetrics and Gynecology, Erciyes University Hospital.

DETAILED DESCRIPTION:
This study was designed to investigate the effect of virtual reality (VR) glasses on pain and anxiety levels experienced by women during gynecological examinations. It was conducted as a randomized controlled experimental study between February and November 2024 at Erciyes University Gevher Nesibe Hospital, Department of Obstetrics and Gynecology.

A total of 126 participants were randomly assigned to intervention and control groups (63 each). Inclusion criteria included women aged between 19 and 49 years, literate, and voluntarily agreeing to participate. Women with gynecological cancer, communication impairments, or visual/auditory disabilities were excluded.

The intervention group received standard gynecological examination procedures along with VR glasses showing immersive nature videos during the examination. The control group underwent the examination without VR intervention. Data collection tools included a Personal Information Form, Pain Beliefs Questionnaire, the Visual Analog Scale (VAS) for pain, and the State-Trait Anxiety Inventory-I (STAI-I) for anxiety. In addition, a Satisfaction Form was applied to the intervention group after the examination.

The aim of the study was to determine whether VR application can reduce perceived pain and anxiety during gynecological procedures. The findings of this study are expected to contribute to non-pharmacological nursing interventions in women's health practices.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 19 and 49 years
* Literate and able to complete the questionnaire
* Agree to participate voluntarily
* Undergoing gynecological examination

Exclusion Criteria:

* Having a diagnosed gynecological cancer
* Hearing or visual impairments
* Cognitive or communication difficulties
* History of psychiatric illness
* Refusal to wear VR glasses

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Change in State Anxiety Score (STAI-I) | Baseline (immediately before the examination) and Post-procedure (within 15 minutes after the examination)
  The State Anxiety Inventory (STAI-I) consists of 20 self-report items that measure how the individual feels at a specific moment. Each item is rated on a 4-point Likert scale: 1 (Not at all) to 4 (Very much so). The scale includes both direct and reverse-scored items. Reverse-scored items include items 1, 2, 5, 8, 10, 11, 16, 19, and 20. The total score is calculated by subtracting the sum of reverse-scored items from the sum of direct items and then adding 50. Total scores range from 20 to 80, with higher scores indicating greater anxiety. The questionnaire will be administered immediately before and 15 minutes after the gynecological examination. The change in scores will be analyzed to evaluate the intervention's effectiveness.
Visual Analog Scale for Pain (VAS) | Post-procedure (within 10 minutes after the gynecological examination)
  The Visual Analog Scale for Pain (VAS) is a widely used unidimensional tool designed to assess subjective pain intensity. It consists of a 10-centimeter horizontal line anchored by two descriptors: "no pain" on the left end and "worst imaginable pain" on the right. Participants will be asked to place a mark along the line that best reflects the intensity of their current pain. The distance (in centimeters) from the left end to the mark will be measured, yielding a score between 0 and 10, with higher scores indicating greater pain intensity. The VAS will be administered once, within 10 minutes following the gynecological examination.

SECONDARY OUTCOMES:
Pain Beliefs Questionnaire - PBQ) | Baseline (within 30 minutes before the gynecological examination)
  The Pain Beliefs Questionnaire (PBQ) will be administered immediately before the gynecological examination to evaluate participants' beliefs about pain.
  The PBQ contains 12 items divided into two subscales:
  Organic Beliefs Subscale (8 items): Items 1, 2, 3, 5, 7, 8, 10, 11
  Psychological Beliefs Subscale (4 items): Items 4, 6, 9, 12
  Each item is rated using a 6-point Likert scale (1 = always, 2 = almost always, 3 = often, 4 = sometimes, 5 = rarely, 6 = never).
  Scores for each subscale will be calculated by averaging the responses of the corresponding items. There is no cutoff point. Higher scores reflect stronger beliefs related to the respective dimension.
  The total score range for each subscale is 1 to 6. Higher scores indicate stronger organic or psychological beliefs about pain.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Bayraktar, PhD, Study Chair — Erciyes University Faculty of Health Sciences
Locations (1):
- Erciyes University Gevher Nesibe Hospital, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy considerations and ethical restrictions imposed by the institutional review board.